CLINICAL TRIAL: NCT02626013
Title: A Multicenter, Prospective Cohort Study to Provide Real-world Evidence on the Effect of Nab-paclitaxel (ABRAXANE®) Treatment on the Clinical Outcomes and Health-related Quality of Life in Patients With Metastatic Breast Cancer in Greece. The 'ABReast' Study.
Brief Title: Real-world Evidence Prospective Study on the Effect of Nab-paclitaxel Treatment on the Clinical Outcomes and HRQoL in Patients With MBC in Greece
Acronym: ABReast
Status: Completed | Type: Observational
Sponsor: Genesis Pharma S.A. (Industry)
Responsible Party: Sponsor
Other Study IDs: NIPMS-GENESIS-ONCO-GRC-001
Record Dates: First submitted 2015-11-25; First posted 2015-12-10 (Estimated); Last update posted 2020-11-30 (Actual); Status verified 2020-11

CONDITIONS: Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This non-interventional study aims at assessing the impact of nab-paclitaxel on the clinical outcomes and the health-related QoL (HRQoL) of this heavily burdened and difficult-to-treat population. Notably, the data generated in the context of this study will serve as complementary evidence to that of the tightly and strictly controlled pre-registration clinical trial setting, which is of essential importance especially in patient populations with diseases of complex and heterogeneous biology, such as breast cancer.

ELIGIBILITY:
Inclusion Criteria:

Patients eligible for inclusion in this study have to meet all of the following criteria:

* Adult patients (18 years and older);
* Patients with a histologically or cytologically confirmed diagnosis of MBC who have failed first-line treatment for metastatic disease and for whom standard, anthracycline containing therapy is not indicated;
* Patients for whom the decision to prescribe therapy with nab-paclitaxel according to the locally approved product's summary of product characteristics (SmPC) has already been taken prior to their enrolment in the study; the assignment of the patient to this therapeutic strategy is not decided in advance by the study protocol but falls within current practice and the prescription of nab-paclitaxel is clearly separated from the physician's decision to include the patient in the current study;
* Patients must be able and willing to provide written informed consent and to comply with the requirements of this study protocol;
* Patients must have signed an informed consent document;
* Patients must be able to read, understand and complete the study specific questionnaire

Exclusion Criteria:

A patient who meets any of the following criteria will be excluded from participation in this study:

* Patients who have initiated treatment with nab-paclitaxel more than 7 days prior to their enrolment into the study;
* Patients that meet any of the contraindications to the administration of the study drug according to the approved SmPC;
* Receipt of any investigational agent within 30 days or 5 half-lives of the investigational agent (whichever is longer) before the commencement of therapy with nab-paclitaxel.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with a histologically or cytologically confirmed diagnosis of MBC who have failed first-line treatment for metastatic disease and for whom standard, anthracycline containing therapy is not indicated
Sampling Method: Probability Sample
Enrollment: 156 (Actual)
Dates: Start 2016-04-12 (Actual); Primary Completion 2018-09-12 (Actual); Study Completion 2018-09-12 (Actual)

PRIMARY OUTCOMES:
Evaluation of the best objective response to nab-paclitaxel treatment in eligible MBC patients as measured from the start of therapy until disease progression, unacceptable toxicity, or termination of study participation | as measured by routine assessments from the start of nab-paclitaxel therapy (at least 6 months post-treatment onset and up to 12 months) until disease progression, occurrence of unacceptable toxicity, or study participation termination
  The proportion of objective responders [patients with either a complete response (CR) or a partial response (PR) as the best objective response] as measured by routine assessments from the start of nab-paclitaxel therapy until disease progression, occurrence of unacceptable toxicity, or study participation termination whichever occurs sooner

CONTACTS AND LOCATIONS:
Overall Officials: Kiki Karvounis, Study Director — GenesisPharma Medical Department
Locations (1):
- Athens, Athens, Greece

REFERENCES:
- [Result] Koumarianou A, Makrantonakis P, Zagouri F, Papadimitriou C, Christopoulou A, Samantas E, Christodoulou C, Psyrri A, Bafaloukos D, Aravantinos G, Papakotoulas P, Baka S, Andreadis C, Alexopoulos A, Bompolaki I, Kampoli Kappa, Liori S, Karvounis K, Ardavanis A. ABREAST: a prospective, real-world study on the effect of nab-paclitaxel treatment on clinical outcomes and quality of life of patients with metastatic breast cancer. Breast Cancer Res Treat. 2020 Jul;182(1):85-96. doi: 10.1007/s10549-020-05677-4. Epub 2020 May 16. PMID 32418045
- See also: Abstract published at Breast Cancer Research & Treatment. Epub 2020 May 16. — https://pubmed.ncbi.nlm.nih.gov/32418045/